CLINICAL TRIAL: NCT05443022
Title: Effect of Photobiomodulation on the Salivary Glands of Patients With Xerostomia and Hyposalivation Induced by the Use of Benzodiazepines - Study Protocol for a Randomized Clinical Trial
Brief Title: Photobiomodulation on the Salivary Glands of Patients With Xerostomia Induced by the Use of Benzodiazepines
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cícero
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The placebo group will have a simulation of application of the laser, with the device turned off. Because it is an infrared light, it is invisible and this will not induce the patient to notice that the device is turned off. In the group that receives the photobiomodulation the device will have its timer turned off, to avoid the perception of sound difference.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Active Comparator): Participants in this group will have their larger salivary glands irradiated with diode laser.
  Interventions: Radiation: Photobiomodulation
- Placebo group (Placebo Comparator): Participants in this group will be subjected to a simulation, where the application protocol will be repeated, but with the laser turned off.
  Interventions: Radiation: Simulation of Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — Participants will receive an application of low intensity light directly in the region of the three pairs of salivary glands. The ArGaAl diode laser, DMC 808nm 4J/point equipment will be used. The parameters that will be used are: Laser Diode ArGaAl, DMC, 808nm, 4J per point, continuously and in contact with the irradiated surface, resulting in irradiance of 3571 mW/cm2, distributed as follows: 6 points in each parotid, 2 points in each sublingual (external) and two in each submandibular (internal), totaling 16 extra oral and 4 intra oral, totaling 20 points. The exposure time will be 40s per point, corresponding to 800s per session and 3600s at the end of the four treatment sessions. The radiant exposure will be 142J/cm2.
  Arms: Photobiomodulation group
Radiation: Simulation of Photobiomodulation — The placebo group will have a simulation of the application of the laser, following the same technique as the active group, but with the device turned off. Because it is an infrared light, it is invisible and this will not induce the patient to notice that the device is turned off.
  Arms: Placebo group

SUMMARY:
Depression is the most common mental illness and antidepressants are in the first line of treatment of depressed patients. This therapeutic class is inevitably associated with side effects and adverse reactions, xerostomia being a symptom that seems to be transverse to them all. Saliva performs multiple functions and plays a vital role in protecting the health of the soft and hard tissues of the oral cavity. Reductions in salivary flow are most often manifested as dry mouth, and this is the subjective complaint called xerostomia. Although xerostomia is the most frequent indication of reduced salivary production, it is not invariably associated with hyposalivation. The user of antidepressant drugs has a number of important systemic and oral complications. Treatment for salivary changes remains unknown, but low-level laser therapy has been shown to be effective in improving salivary flow in patients with xerostomia due to diabetes, Sjogren's syndrome, chemotherapy and radiotherapy for head, neck and lung cancer. This randomized controlled trial aims to evaluate oral symptoms related to salivary gland function and mucosal condition of depressed patients, as well as the effects of photobiomodulation on salivary flow. Sixty patients will be included in the protocol, after signing the Informed Consent Form. They will undergo anamnesis, physical evaluation and oral health self-perception questionnaires and symptoms related to salivary gland function and then will be divided into two groups: Photobiomodulation (PBM) (n=30); will have their larger salivary glands irradiated with Diode laser (808nm, 4J per point, 40s) and placebo (PCB) (n=30), which will be subjected to a simulation, where the application protocol will be repeated, but with the laser off. Previous and post treatment sialometries will be performed to compare saliva volume. Biochemical analysis, in which total protein and calcium will be measured, will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Participants in good general health, but who have depression with regular use of benzodiazepines;
* Complaints of xerostomia or hyposalivation;
* Over 18 years of age;
* Be able to understand and sign the Informed Consent Form.

Exclusion Criteria:

* Participants who present current acute systemic infectious conditions;
* Chronic kidney disease;
* Diabetics;
* Participants with a history of mental disorders other than depression and anxiety;
* Participants without conditions for dental treatment in the month of referral to the dental service;
* Hemodynamic instability;
* Signs and symptoms related to the cardiovascular systems;
* Acute systemic infectious processes;
* Acute cardiovascular disease;
* Those with any type of photosensitivity;
* Neoplasms in the region of glands;
* Under 18 years of age;
* Pregnant or lactating women;
* Participants with xerostomia not induced by anxiolytics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Sialometry (measurement of the amount of produced saliva before and after treatment) | Baseline and immediately after treatment.
  The patient will be instructed to keep the head forward allowing all saliva to passively pass through the collection tube, resting on the lower lip, for five minutes. In the last second, the patient will be instructed to spit out all the accumulated saliva in the collection tube. The amount of saliva and foam will be evaluated and properly recorded. Then, the dimethicone (removal of the air bubbles) will be used to obtain the final result. At the end of the photobiomodulation session, a sample of saliva will be collected to be compared to the initial sample. The measurement will be made as follows: milliliters of saliva produced per minute. For stimulate sialometry, a sialogogue will be used. The quantity will be classified as follows: Production of normal saliva: 1.5 to 3.0 ml/minute; Light hyposalivation: from 1.05 to 1.45 ml/minute; Moderate hyposalivation: 0.55 to 1.0 ml/minute; Severe hyposalivation: from 0.05 to 0.50 ml/minute; Sialorrhea: above 3.0 ml/min.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil